CLINICAL TRIAL: NCT04494269
Title: An Open-label, Multi-center, Single-dose, Parallel-group Study to Evaluate Pharmacokinetics and Safety of Tegoprazan in Subjects With Hepatic Impairment and Healthy Controls
Brief Title: A Study to Evaluate Pharmacokinetics and Safety of Tegoprazan in Subjects With Hepatic Impairment and Healthy Controls
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN_APA_116
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-07

CONDITIONS: Hepatic Impairment; Healthy
MeSH Terms: interventions — tegoprazan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subjects with normal hepatic function (Active Comparator): Single dose of Tegoprazan 50mg
  Interventions: Drug: Tegoprazan 50mg
- Subjects with mild hepatic impairment (Experimental): Single dose of Tegoprazan 50mg
  Interventions: Drug: Tegoprazan 50mg
- Subjects with moderate hepatic impairment (Experimental): Single dose of Tegoprazan 50mg
  Interventions: Drug: Tegoprazan 50mg
- Subjects with severe hepatic impairment (Experimental): Single dose of Tegoprazan 50mg
  Interventions: Drug: Tegoprazan 50mg

INTERVENTIONS:
Drug: Tegoprazan 50mg — Oral administration once daily
  Other Names: K-CAB

SUMMARY:
The main purpose of this study is to compare the pharmacokinetic and safety of tegoprazan following single oral dose in subjects with hepatic impairment versus healthy control.

DETAILED DESCRIPTION:
[Pharmacokinetic Assessment]

* Measurements

  - Tegoprazan and desmethyl tegoprazan (M1) in blood and urine
* Endpoints

  * Primary endpoints: AUClast and Cmax of tegoprazan and M1
  * Secondary endpoints: CL/F, t1/2, AUCinf, and fu of tegoprazan; CLrenal and Ae of tegoprazan and M1

[Safety Assessment]

* Adverse events (AEs)
* Clinical laboratory tests
* Vital sign
* Physical examination
* Electrocardiogram (ECG)

ELIGIBILITY:
[Healthy Control Group]

Inclusion Criteria:

* Subjects aged 19 to 70(inclusive) years at the time of signing the informed consent form.
* Subjects with a body weight of ≥ 50 kg and ≤ 90 kg at screening.
* Subjects with AST, ALT, and ALP levels of ≤ 1.5 × upper limit of the normal reference range (ULN) with total bilirubin < 2 mg/dL and PT (INR) < 1.7 at screening.
* Subjects who have no chronic disease or any congenital disease within the last 5 years and no pathological symptoms or findings as a result of an internal examination
* Subjects who provide voluntary written informed consent to study participation after being informed of detailed explanation and fully understanding study objectives, procedures and characteristics of the investigational product(IP).

Exclusion Criteria:

* Subjects who show symptoms of acute disease at the time of screening.
* Subjects with any clinically significant disease related to ongoing cardiovascular problem, respiratory system, kidney, endocrine system, hematologic, central nervous system, mental health disorder, or malignant tumor.
* Subjects with history or current evidence of gastrointestinal or hepatobiliary disease which may affect PK evaluation of the IP.
* Subjects with history or current evidence of clinically significant hypersensitivity to drugs containing any ingredient of proton pump inhibitors or potassium-competitive acid blockers and other drugs (such as aspirin and antibiotics).
* Subjects with systolic blood pressure (BP) of < 90 mmHg or > 160 mmHg, or diastolic BP of < 50 mmHg or > 100 mmHg at screening.
* Subjects who have received medication or food which may significantly affect absorption, distribution, metabolism, or elimination of study drug within 7 days prior to scheduled study treatment.
* Subjects who have participated in any other clinical study or bioequivalence study and received investigational agent within 180 days prior to scheduled study treatment.
* Subjects who have donated whole blood within 60 days prior to the scheduled study treatment, or has donated blood components or received transfusion within 30 days prior to scheduled study treatment.
* Subjects who are unable to use a medically acceptable contraceptive method throughout the study.
* Subjects who are determined ineligible for study participation by the investigator for other reasons.

[Subjects with Hepatic Impairment]

Inclusion Criteria:

* Subjects with chronic liver disease who meet any of the followings:

  * Chronic Hepatitis B;
  * Chronic Hepatitis C;
  * Alcoholic liver disease;
  * Non-alcoholic fatty liver disease; or
  * Liver fibrosis and cirrhosis.
* Subjects aged 19 to 70 years (inclusive) at the time of signing the informed consent form.
* Subjects with body weight of ≥ 50 kg and ≤ 90 kg with a BMI of ≥ 18.0 kg/m2 and ≤ 30 kg/m2 at screening.
* Subjects who meet any of following criteria:

  * AST, ALT, or ALP level > 1.5 × ULN at screening;
  * Total bilirubin ≥ 2 mg/dL at screening; or
  * PT (INR) ≥ 1.7 at screening.
* Subjects who provide voluntary written informed consent to study participation after being informed of detailed explanation and fully understanding study objectives, procedures and characteristics of the IP.

Exclusion Criteria:

* Subjects who show symptoms of acute disease at the time of screening.
* Subjects with any clinically significant disease related to ongoing cardiovascular problem, respiratory system, kidney, endocrine system, hematologic, central nervous system, mental health disorder, or malignant tumor.
* Subjects with a history or current evidence of gastrointestinal disease which may affect PK evaluation for the IP.
* Subjects who have clinical changes to an estimated level that may affect PK evaluation of the study drug within 30 days prior to the scheduled dosing date.
* Changes in existing medications including dosage regimen within 30 days prior to the scheduled dosing date.
* Subjects with prior history or current evidence of clinically significant hypersensitivity to drugs containing any ingredient of proton pump inhibitors or potassium-competitive acid blockers and other drugs (such as aspirin and antibiotics).
* Systolic BP of < 90 mmHg or > 160 mmHg, or diastolic BP of < 50 mmHg or > 100 mmHg at screening.
* Any concomitant medications or foods which may significantly affect absorption, distribution, metabolism, or elimination of the study drug within 7 days prior to the scheduled dosing date.
* Subjects who have participated in any other clinical study or bioequivalence study and received investigational agent within 180 days prior to scheduled study treatment.
* Subjects who have donated whole blood within 60 days prior to the scheduled dosing date, or have donated blood components or received transfusion within 30 days prior to the scheduled dosing date.
* Subjects who are unable to use medically acceptable contraceptive methods throughout the study.
* Subjects who are determined to be ineligible for study participation by the investigator for other reasons.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment | Up to 48 hours
  AUClast of tegoprazan and M1
Pharmacokinetic Assessment | Up to 48 hours
  Cmax of tegoprazan and M1

SECONDARY OUTCOMES:
Pharmacokinetic Assessment | Up to 48 hours
  CL/F of tegoprazan
Pharmacokinetic Assessment | Up to 48 hours
  t½ of tegoprazan
Pharmacokinetic Assessment | Up to 48 hours
  AUCinf of tegoprazan
Pharmacokinetic Assessment | Up to 48 hours
  fu of tegoprazan
Pharmacokinetic Assessment | Up to 48 hours
  CLrenal of tegoprazan and M1
Pharmacokinetic Assessment | Up to 48 hours
  Ae of tegoprazan and M1

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Ryul Kim, MD, PhD, Study Chair — Samsung Medical Center; Yang-Won Min, MD, PhD, Principal Investigator — Samsung Medical Center; Dong-Seong Shin, MD, PhD, Principal Investigator — Gachon University Gil Medical Center; Eon-Hye Kim, MD, PhD, Principal Investigator — CHA Bundang Medical Center
Locations (3):
- South Korea (3):
  - Gachon University Gil Medical Center, Incheon
  - CHA Bundang Medical Center, Seongnam-si
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Kim A, Shin D, Seo Y, Kang D, Min YW, Kim IH, Kim J. Phase I Study to Evaluate the Effect of Hepatic Impairment on Pharmacokinetics and Safety of Tegoprazan, a Potassium Competitive Acid Blocker. Adv Ther. 2025 Mar;42(3):1570-1581. doi: 10.1007/s12325-025-03127-5. Epub 2025 Feb 11. PMID 39932678